CLINICAL TRIAL: NCT00052962
Title: A Prospective Random Assignment Trial to Study Operative Debulking and Systemic Chemotherapy With or Without Intra-and Peri-Operative Intraperitoneal Chemotherapy for Subjects With Peritoneal Carcinomatosis From Low Grade Gastrointestinal Adenocarcinoma
Brief Title: Debulking and Chemotherapy With or Without Intraperitoneal Chemotherapy to Treat Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marybeth Hughes, Marybeth Hughes, M.D., National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030085; 03-C-0085; NCT00056108 (obsolete NCT alias)
Record Dates: First submitted 2003-01-26; First posted 2003-01-27 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Appendiceal Cancer; Regional Therapy; Carcinomatosis; Hyperthermia
MeSH Terms: conditions — Gastrointestinal Neoplasms; Appendiceal Neoplasms; Carcinoma; Hyperthermia | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Surgery + post op chemotherapy (Other): * Cytoreductive surgery - patients will undergo a laparotomy, surgical incision in the abdomen to assess the peritoneal cavity, with cytoreductive surgery, or tumor debulking to reduce tumor size.
  * Post operative chemotherapy: systemic oxaliplatin, leucovorin and infusional 5-fluorouracil (5-FU), every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles {16 weeks total}.
  Interventions: Procedure: Cytoreductive surgery
- Arm 2 Surgery + HIPEC (Other): Arm 2 Surgery + Continuous hyperthermic peritoneal perfusion (CHPP/HIPEC) + post op dwell + post op chemotherapy
  * Cytoreductive surgery - patients will undergo a laparotomy, surgical incision in the abdomen to assess the peritoneal cavity, with cytoreductive surgery, or tumor debulking to reduce tumor size.
  * followed by continuous hyperthermic peritoneal perfusion (HIPEC) with 250 mg/m^2 cisplatin
  * post operative dwell chemotherapy given once between post op day 7 and 12: 5-fluorouracil (5FU) 800 mg/m^2 and paclitaxel 125 mg/m^2
  * post operative chemotherapy: systemic oxaliplatin, leucovorin and infusional 5-FU, every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles {16 weeks total}.
  Interventions: Procedure: Cytoreductive surgery; Procedure: Continuous hyperthermic peritoneal perfusion (HIPEC/CHPP)

INTERVENTIONS:
Procedure: Cytoreductive surgery — Patients will undergo a laparotomy, surgical incision in the abdomen to assess the peritoneal cavity with cytoreductive surgery or tumor debulking, to reduce tumor size.
  Drug: Post operative chemotherapy: systemic oxaliplatin 85 mg/m^2 on day 1 only, leucovorin 200 mg/M^2/day on day 1, 2, 15, and 16, and infusional 5-flurouracil (5-FU) 800 mg/m^2 on day 8, every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles { 16 weeks total}.
Procedure: Continuous hyperthermic peritoneal perfusion (HIPEC/CHPP) — Patients will undergo a laparotomy, surgical incision in the abdomen to assess the peritoneal cavity with cytoreductive surgery or tumor debulking, to reduce tumor size.
  Followed by continuous hyperthermic peritoneal perfusion (HIPEC) with 250 mg/m^2 cisplatin. Post operative dwell chemotherapy given once between post op day 7 and 12: 5-fluororacil (5-FU) 800 mg/m^2 and paclitaxel 125 mg/m^2.
  Drug: Post operative chemotherapy: systemic oxaliplatin 85 mg/m^2 on day 1 only, leucovorin 200 mg/M^2/day on day 1, 2, 15, and 16, and infusional 5-flurouracil (5-FU) 800 mg/m^2 on day 8, every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles { 16 weeks total}.
  Arms: Arm 2 Surgery + HIPEC

SUMMARY:
This study will determine which of the two following treatment regimens provides greater benefit to patients with peritoneal carcinomatosis (gastrointestinal cancer that has spread throughout the abdomen):

* Surgical removal of tumors plus heated chemotherapy during surgery, followed by one dose of chemotherapy 7 to 12 days after surgery, followed 3 weeks later by 4 months of chemotherapy; or
* Surgical removal of tumors followed by 4 months of chemotherapy, starting 1 month after surgery.

Patients 18 years of age and older with peritoneal carcinomatosis may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood tests; chest X-ray and computed tomography (CT) scans; review of pathology slides; electrocardiogram (EKG), bone scan, and brain magnetic resonance imaging (MRI), as needed; and laparotomy. Laparatomy is a surgical procedure in which an incision is made in the abdomen to look at the amount and location of tumors in the abdominal cavity. Patients whose surgery reveals that the tumors cannot be removed are taken off study. Those eligible for the study have their tumors removed during this screening laparotomy as part of the study procedure, as follows:

All participants undergo laparotomy and removal of as much tumor as possible, as described above. Patients are then randomly assigned to one of two treatment groups:

* Group 1 - During laparotomy, after tumor removal, patients receive continuous hyperthermic peritoneal perfusion (CHPP) with the anti-cancer drug cisplatin. For CHPP, the cisplatin solution is heated and delivered to the abdomen through a catheter (plastic tube), washed through the abdomen for 90 minutes, and then drained out of the body through another catheter. At the close of surgery, a small catheter, called a Tenckhoff catheter, is left in the abdomen and brought out through the skin. Between days 7 and 12 after surgery, one dose of fluorouracil and paclitaxel chemotherapy is delivered through this catheter. The catheter is removed following complete recovery from surgery and the patient is discharged from the hospital. Four to 6 weeks after the surgery, patients have CT scans of the chest, pelvis, and abdomen, and then begin intravenous (IV, through a vein) chemotherapy with oxaliplatin, 5-fluorouracil (5-FU), and leucovorin. The chemotherapy is given in 4-week courses as follows: oxaliplatin on day 1, infused over 2 hours through a vein in the arm or neck; leucovorin on days 1 and 2, infused over 2 hours, followed by 5-fluorouracil over 22 hours; leucovorin and 5-FU repeated two weeks later on days 15 and 16. This regimen is repeated two weeks later. Between each week of chemotherapy is a week break. A course of chemotherapy consists of 28 days (two weeks of chemotherapy and two 1-week breaks). Patients may receive up to four courses (total of 16 weeks) unless their disease progresses or they cannot tolerate further doses. Doses of the chemotherapy can be reduced if the side effects are too severe.
* Group 2 - Patients follow the same procedure as those in Group 1 for laparotomy, CT imaging, and IV chemotherapy with oxaliplatin, 5-fluorouracil, and leucovorin. They do not receive CHPP or chemotherapy into the abdomen.

All patients undergo repeat imaging tests six weeks after surgery and at the conclusion of the intravenous (IV) chemotherapy. They return for a physical examination and CT scans every three months for the first year, every four months for the next two years, and then every six months for up to five years after treatment. They are also asked to complete quality of life questionnaires before and after surgery, at the completion of chemotherapy, and at every follow-up visit.

DETAILED DESCRIPTION:
Patients with low-grade gastrointestinal adenocarcinoma and peritoneal carcinomatosis will undergo laparotomy and tumor debulking. Patients will be randomized at completion of tumor debulking to receive continuous hyperthermic peritoneal perfusion (HIPEC,formerly CHPP) with 250 mg/m^2 cisplatin and an intraperitoneal dwell of 5-fluorouracil 800 mg/m^2 and paclitaxel 125 mg/m^2 once between postoperative day 7 and 12. All patients will receive systemic oxaliplatin, leucovorin and infusional 5-FU, every other week of every four weeks starting 4 to 6 weeks after operation and continuing for four cycles. The major endpoint is time to intraperitoneal tumor progression and survival in patients stratified based on history of previous treatment with systemic chemotherapy (yes vs. no), history of prior debulking surgery; and ability to optimally vs. suboptimally debulk intraperitoneal tumor burden.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. The patient must have histologically or cytologically proven peritoneal carcinomatosis from low-grade mucinous adenocarcinoma of the gastrointestinal tract. Patients with no tissue for examination may undergo percutaneous needle aspiration under computed tomography (CT) or ultrasound guidance as clinically indicated or a laparotomy with biopsy if a tumor grade cannot be determined on other available material.
  2. Radiologic workup must demonstrate that there is no imageable disease outside of the peritoneal cavity.
  3. Radiologic workup or prior abdominal exploration must show abnormalities consistent with disease which can be debulked to a residual size of less than 1 cm in diameter per tumor deposit in the judgement of the investigators.
  4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2 on study entry and on the day prior to planned treatment.
  5. Patients must have a minimum expected duration of survival of greater than 16 weeks.
  6. Patients must have recovered from any severe toxicity from all prior chemotherapy, immunotherapy or radiotherapy except as outlined in appendix 1 of the protocol and be at least 30 days past the date of their last treatment.
  7. Patients must have a serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within 5 times the upper limit of normal and a total serum bilirubin of less than 3 times the upper limit of normal, both of which define the upper limit of grade 2 treatment related toxicities..
  8. Patients must have a absolute neutrophil count (ANC) greater than 1,500/microliter.
  9. Patients must be age greater than or equal to 18 years.

EXCLUSION CRITERIA:

1. Patients will be excluded if they have concomitant medical problems that would place them at unacceptable risk for a major surgical procedure.

   1. Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g. age greater than 65, and a history of hypertension, first degree relative with atherosclerotic coronary artery evaluation and will not be eligible if they demonstrate significant irreversible ischemia on a stress thallium study or an ejection fraction of less than 40%.
   2. Patients who have shortness of breath with minimal exertion or who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing and will not be eligible if their forced expiratory volume 1 (FEV1) is less than 1.2 liters or their maximum voluntary ventilation is less than 50% of expected.
2. Patients who have a neurological toxicity of Grade 3 or greater will be excluded because of the potential neurotoxicity associated with platinum and paclitaxel therapy.
3. Patients will be ineligible if they have a serum creatinine of greater than 1.5 mg/dL unless the measured creatinine clearance is greater than 60mL/min/1.73m^2.
4. Patients will be ineligible if platelets are less than 75, 000/mm^3.
5. Patients who have failed previous intraperitoneal chemotherapy will be ineligible.
6. Pregnant women or women who are breast-feeding will be ineligible.
7. Patients less than 30 kg will be ineligible.
8. Patients who have undergone two or more operative procedures to debulk disease, have received 2 or more regimens of systemic chemotherapy, or any previous continuous hyperthermic peritoneal perfusion (CHPP) therapy will be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Douillard JY, Cunningham D, Roth AD, Navarro M, James RD, Karasek P, Jandik P, Iveson T, Carmichael J, Alakl M, Gruia G, Awad L, Rougier P. Irinotecan combined with fluorouracil compared with fluorouracil alone as first-line treatment for metastatic colorectal cancer: a multicentre randomised trial. Lancet. 2000 Mar 25;355(9209):1041-7. doi: 10.1016/s0140-6736(00)02034-1. PMID 10744089
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2003-C-0085.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Surgery + Post op Chemotherapy: * Cytoreductive surgery
  * Post operative chemotherapy: systemic oxaliplatin, leucovorin and infusional 5-fluorouracil (5-FU), every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles {16 weeks total}.
- Arm 2 Surgery + CHPP: Arm 2 Surgery + Continuous hyperthermic peritoneal perfusion (CHPP) + post op dwell + post op chemotherapy
  * Cytoreductive surgery
  * continuous hyperthermic peritoneal perfusion (CHPP) with 250 mg/m^2 cisplatin
  * post operative dwell chemotherapy given once between post op day 7 and 12: 5-fluorouracil (5FU) 800 mg/m^2 and paclitaxel 125 mg/m^2
  * post operative chemotherapy: systemic oxaliplatin, leucovorin and infusional 5-FU, every other week of every four weeks (two weeks per month) starting 4 to 6 weeks after operation and continuing for four cycles {16 weeks total}.
Period: Overall Study
Arm/Group | Arm 1 Surgery + Post op Chemotherapy | Arm 2 Surgery + CHPP
Started | 13 | 17
Completed | 12 | 15
Not Completed | 1 | 2
Not completed — Not evaluable | 0 | 2
Not completed — Not randomized/not evaluable | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Surgery + Post op Chemotherapy | Arm 2 Surgery + CHPP | Total
Number analyzed (Participants) | 13 | 17 | 30
Age Categorical [Number; unit: Participants] — Two subject's were not evaluable, and/or information is not known for Arm 2.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 15 | 26
    >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] — Mean values were not calculated for all participants who started the study because one participant was not randomized/not evaluable, two were not evaluable, and/or information is not known.
  years | 51.08 (15.58) | 48.64 (11.21) | 50.55 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 16 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 10 | 13 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: CHPP is administered as a heated cisplatin solution delivered to the abdomen through a catheter (plastic tube), washed through the abdomen for 90 minutes, and then drained out of the body through another catheter.
  Progression is defined as imageable tumor nodules or increasing ascites persistent on two serial computed tomography (CT) scans.
Time Frame: 2003-2008
Population: Study was closed July 2008 because the PI left the institution, thus the objective was not met.
Arm/Group | Arm 1 Surgery + Post op Chemotherapy | Arm 2 Surgery + CHPP
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With an Adverse Event
Description: Here is the number of participants with an adverse event. For a detailed list of adverse events see the adverse event module.
Time Frame: 2003-2008
Population: Three participants were not included in the analysis because one participant was not randomized/not evaluable, two were not evaluable, and/or information is not known.
Measure: Number; unit: Participants
Arm/Group | Arm 1 Surgery + Post op Chemotherapy | Arm 2 Surgery + CHPP
Number analyzed (Participants) | 13 | 14
Participants | 7 | 6

ADVERSE EVENTS:
Description: Three participants were no included in the assessment because one participant was not randomized/not evaluable, two were not evaluable, and/or information is not known.
Arm/Group | Arm 1 Surgery + Post op Chemotherapy | Arm 2 Surgery + CHPP
Serious Adverse Events (participants affected / at risk) | 5/13 | 6/14
Other Adverse Events (participants affected / at risk) | 2/13 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Surgery + Post op Chemotherapy (N=13) | Arm 2 Surgery + CHPP (N=14)
Ileus, wound infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lipase gr (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fistula intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Partial small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Post-op ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound infection (superficial) (Infections and infestations) | 1 (1) | 0 (0)
AST (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bowel perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion/non-malignant (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abd pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bilateral pleural effusion, bibasilar atelectasis, pelvic fluid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ALT/AST (Hepatobiliary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Surgery + Post op Chemotherapy (N=13) | Arm 2 Surgery + CHPP (N=14)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
SVT (Cardiac disorders) | 1 (1) | 0 (0)
UTI: pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion post op (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No